CLINICAL TRIAL: NCT01791179
Title: Carolina Alcohol and Drug Resources
Acronym: CADRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00042125; 1H79TI024350-01 (NIH)
Record Dates: First submitted 2013-02-12; First posted 2013-02-13 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Substance Abuse Treatment Group (Experimental)
  Interventions: Behavioral: Comprehensive substance abuse services

INTERVENTIONS:
Behavioral: Comprehensive substance abuse services

SUMMARY:
Substance abuse is highly prevalent among individuals with HIV and associated with negative outcomes including poorer medication adherence and HIV risk behavior. The primary aim of this project is to address substance abuse among individuals with or at high-risk for HIV by enhancing and expanding the substance abuse services provided in the formerly Substance Abuse and Mental Health Services Administration (SAMHSA) funded Carolinas Alcohol and Drug Expansion Team (CADET) program, which offered comprehensive substance abuse care for individuals with HIV living primarily in the Durham NC area. Services will be enhanced by adding peer outreach and navigation services to improve treatment engagement and participation and expanded to replicate the enhanced CADET service model in Charlotte NC.

The target population for this project is minority individuals, primarily African-Americans, with HIV or at high-risk for HIV with a particular focus on minority men who have sex with men (MSM)s. The program will provide up to 18 months of comprehensive services for approximately 315 individuals and will include: 1) peer outreach to facilitate and enhance treatment engagement 2) individual and group substance abuse treatment using evidence-based models 3) ongoing recovery groups for individuals who have completed the intensive substance abuse treatment phase and 4) linkage to needed services such as case management, psychiatric care, and HIV/Hepatitis medical care. We will also target HIV and Hepatitis C testing and treatment services for minority MSM of unknown HIV status to increase access and utilization of substance use services and identify HIV and Hepatitis status.

The study evaluation will involve analysis of participant survey data gathered at baseline, 6, 12, 18 months of study participation to determine the effect of the comprehensive substance abuse care services on outcomes for individuals with HIV including substance use, mental health, HIV treatment adherence, HIV risk behavior, and access and utilization of HIV services. The study will also determine the effect of the comprehensive substance use program on substance abuse, mental health, and risk behavior outcomes for minority MSM who are not HIV-positive.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive or minority MSM
* substance abuse
* 18 or over

Exclusion Criteria:

* Under 18
* cognitive impairment that would preclude participation in substance abuse treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Change in substance use | 12 months
  Substance use information will be collected at baseline, 6, and 12 months through surveys using standardized substance use measures including the Addiction Severity Index (ASI).

SECONDARY OUTCOMES:
Change in medication adherence | 12 months
  HIV medication adherence data will be collected at baseline, 6, and 12 months through surveys using standardized adherence measures in the visual analog scale and CASE adherence measure.

CONTACTS AND LOCATIONS:
Overall Officials: Susan S. Reif, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

REFERENCES:
- See also: Related Info — http://chpir.org